CLINICAL TRIAL: NCT02087163
Title: The Use of Clear Aligners With Movement Enhancement Techniques
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Align Technology, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CSP-700007-00
Record Dates: First submitted 2014-02-28; First posted 2014-03-14 (Estimated); Results first posted 2019-04-24 (Actual); Last update posted 2020-01-31 (Actual); Status verified 2020-01

CONDITIONS: Malocclusion
MeSH Terms: conditions — Malocclusion | interventions — Orthodontic Appliances, Removable

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Movement Enhancement Technique (Experimental): Movement Enhancement Technique Clear Aligner
  Interventions: Device: Movement Enhancement Technique; Device: Clear Aligner

INTERVENTIONS:
Device: Movement Enhancement Technique — Conventional Orthodontic treatment
Device: Clear Aligner — Orthodontic treatment with Clear Aligner

SUMMARY:
The purpose of this study is to use clear aligners to measure tooth movement and length of treatment.

DETAILED DESCRIPTION:
Orthodontic tooth movement is the result of a force applied to the crown of a tooth and the biological remodeling of the gum and bony tissues.

ELIGIBILITY:
Inclusion Criteria:

* Require Orthodontic Treatment
* Have a permanent dentition
* No craniofacial anomaly present
* No past and present signs and symptoms of periodontal disease
* No significant medical history or medication that would adversely affect the development or structure of the teeth and jaws and any subsequent tooth movement
* No previous orthodontic or orthopaedic relapse
* No history of trauma, bruxism or parafunction
* 16- 46 years old, inclusive
* No skeletal jaw discrepancy
* Angle Class I or Class II molar and canine relationship
* Crowding of at least 4mm per arch
* No osteoporosis drugs

Exclusion Criteria:

* Subjects who do not fulfill all inclusion criteria requirements

Ages: 16 Years to 46 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 90 (Actual)
Dates: Start 2014-02; Primary Completion 2018-12 (Actual); Study Completion 2019-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Chenin, Principal Investigator; Kottemann, Principal Investigator; Mariani, Principal Investigator
Locations (1):
- Align Technology, Inc., San Jose, California, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Movement Enhancement Technique
Started | 90
Completed | 73
Not Completed | 17

BASELINE CHARACTERISTICS:
Arm/Group | Movement Enhancement Technique
Number analyzed (Participants) | 90
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 90
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 70
  Male | 20
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 90

OUTCOME MEASURES:

1. Primary Outcome: Tooth Movement Change
Description: Participants will be followed for the duration of orthodontic treatment, an expected average of 78 weeks. Tooth movement change will be measured as the number of millimeters of tooth movement per aligner.
Time Frame: Baseline and end of treatment, an average of 78 weeks
Population: all completed subjects
Measure: Mean (95% Confidence Interval); unit: millimeters
Arm/Group | Movement Enhancement Technique
Number analyzed (Participants) | 73
millimeters | 0.363 [-0.22 to 0.45]

2. Secondary Outcome: Length of Treatment Change
Description: Participants will be followed for the duration of orthodontic treatment, an expected average of 78 weeks. Length of treatment change will be measured as the number of weeks of movement per aligner.
Time Frame: Baseline and end of treatment, an average of 78 weeks
Population: all completed subjects
Measure: Mean (95% Confidence Interval); unit: days
Arm/Group | Movement Enhancement Technique
Number analyzed (Participants) | 73
days | 342 [-37.08 to 441.27]

ADVERSE EVENTS:
Time Frame: baseline until end of treatment, an average of 78 weeks
Description: An adverse event (AE) is any unwanted dental occurrence in a clinical investigation subject whether or not the AE is suspected of having a causal relationship with study treatment. Pre-existing events, which increase in frequency or severity or change in nature during or as a consequence of use of an appliance clinical trials, will also be considered as adverse events.
Arm/Group | Movement Enhancement Technique
All-Cause Mortality (participants affected / at risk) | 0/90
Serious Adverse Events (participants affected / at risk) | 0/90
Other Adverse Events (participants affected / at risk) | 0/90

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-01-09): https://cdn.clinicaltrials.gov/large-docs/63/NCT02087163/Prot_SAP_000.pdf